CLINICAL TRIAL: NCT04487847
Title: 18F-PSMA-1007 PET to Detect Primary Prostate Cancer: a Comparative Study With mpMRI and Correlation to Histopathology
Brief Title: 18F-PSMA-1007 PET Imaging to Detect Primary Prostate Cancer
Acronym: PICture
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ABX advanced biochemical compounds GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL73559.091.20
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Staging; PET imaging; PSMA-1007; mpMRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Explorative study of 18F-PSMA-1007 PET to detect prostate cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PIRADS 1-2 (Experimental): 25 patients with PIRADS 1-2 (probably benign) on mpMRI
  Interventions: Diagnostic Test: 18F-PSMA-1007 PET/CT
- PIRADS 3 (Experimental): 25 patients with PIRADS 3 (equivocal scan) on mpMRI
  Interventions: Diagnostic Test: 18F-PSMA-1007 PET/CT
- PIRADS 4-5 (Experimental): 25 patients with PIRADS 4-5 (probably malignant) on mpMRI
  Interventions: Diagnostic Test: 18F-PSMA-1007 PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-PSMA-1007 PET/CT — 18F-PSMA-1007 PET/CT

SUMMARY:
To study the added value of 18F-PSMA-1007 PET to mpMRI in the detection of local prostate cancer lesions.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the second most common diagnosed malignancy in males worldwide, with over 1.2 million new patients diagnosed every year. Since the introduction of prostate-specific antigen (PSA) the primary diagnosis consisted of histologic confirmation by transrectal ultrasound (TRUS) systematic biopsies. However, in recent years this has changed into performing multi-parametric MR imaging (mpMRI) prior to prostate biopsy.

MpMRI has proven to be a valuable tool to avoid unnecessary prostate biopsies and prevent over-treatment of low-grade PCa, while maintaining equal or higher detection rates of high-grade PCa. Prostate MRI is evaluated using the Prostate Imaging-Reporting and Data System (PIRADS). Lesions are given a category score, from 1 (high-grade PCa is unlikely to be present) to 5 (presence of high-grade PCa is highly likely). A PIRADS 3 is an equivocal scan. Nonetheless, mpMRI has room for improvement as its specificity for high-grade tumors is only 73% and local staging is limited with mpMRI. Also, the mpMRI is frequently unclear as 4-39% of detected lesions are classified as PIRADS 3.

Prostate-specific membrane antigen receptor (PSMA) is highly overexpressed by 95% of the prostate cancer cells and seem to positively correlate to aggressiveness of the tumor. PSMA-positron emission tomography (PET) uses this feature by visualizing PSMA expressing prostate tumors. Currently, the PSMA-PET is generally used to detect recurrences or metastases. However, there is an increasing interest for PSMA-PET scans in patients with a primary diagnosis of PCa for staging purposes. Yet, there is no published data on the role of PSMA-PET on PCa prior to biopsy in comparison to the detection rate of mpMRI and histopathology.

This study aims to investigate the added value of a 18F-PSMA-PET to mpMRI in the detection of local prostate cancer lesions.

75 patients with the suspicion on prostate cancer (e.g. elevated PSA and/or abnormal digital rectal exam) will receive a 18F-PSMA-1007 PET following mpMRI. 25 patients with PIRADS 1-2 (probably benign disease), 25 patients with PIRADS 3 (equivocal disease) and 25 patients with PIRADS 4-5 (highly suspicious for malignancy) will be included in this study.

If either the mpMRI or 18F-PSMA-1007 PET shows a potential malignant lesion, a (target) biopsy will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion for PCa (e.g. elevated PSA, suspicious rectal examination)
* Males ≥ 18 years
* ECOG 0-1
* Signed informed consent

Exclusion Criteria:

* Prostate biopsy in the last 6 months
* History of prostate cancer
* Second active malignancy
* Any prior surgery in the pelvic area that might interfere with the scans (e.g. hip replacement surgery)
* Any medical condition that in the opinion of the investigator will affect patients' clinical status when participating in this trial.
* Contra-indications for mpMRI or PET: claustrophobia or inability to lay still for the duration of the exam.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 75 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Compare mpMRI,18F-PSMA-1007 PET and histopathology. | 30 days
  Within each of the three PIRADS groups (1-2, 3, 4-5) the fraction of patients in which the diagnosis based on mpMRI and 18F-PSMA-1007 PET differ is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH. Diagnostic Performance of Prostate Imaging Reporting and Data System Version 2 for Detection of Prostate Cancer: A Systematic Review and Diagnostic Meta-analysis. Eur Urol. 2017 Aug;72(2):177-188. doi: 10.1016/j.eururo.2017.01.042. Epub 2017 Feb 11. PMID 28196723
- [Result] Barentsz JO, Weinreb JC, Verma S, Thoeny HC, Tempany CM, Shtern F, Padhani AR, Margolis D, Macura KJ, Haider MA, Cornud F, Choyke PL. Synopsis of the PI-RADS v2 Guidelines for Multiparametric Prostate Magnetic Resonance Imaging and Recommendations for Use. Eur Urol. 2016 Jan;69(1):41-9. doi: 10.1016/j.eururo.2015.08.038. Epub 2015 Sep 8. No abstract available. PMID 26361169
- [Result] de Rooij M, Hamoen EH, Witjes JA, Barentsz JO, Rovers MM. Accuracy of Magnetic Resonance Imaging for Local Staging of Prostate Cancer: A Diagnostic Meta-analysis. Eur Urol. 2016 Aug;70(2):233-45. doi: 10.1016/j.eururo.2015.07.029. Epub 2015 Jul 26. PMID 26215604
- [Result] van der Leest M, Cornel E, Israel B, Hendriks R, Padhani AR, Hoogenboom M, Zamecnik P, Bakker D, Setiasti AY, Veltman J, van den Hout H, van der Lelij H, van Oort I, Klaver S, Debruyne F, Sedelaar M, Hannink G, Rovers M, Hulsbergen-van de Kaa C, Barentsz JO. Head-to-head Comparison of Transrectal Ultrasound-guided Prostate Biopsy Versus Multiparametric Prostate Resonance Imaging with Subsequent Magnetic Resonance-guided Biopsy in Biopsy-naive Men with Elevated Prostate-specific Antigen: A Large Prospective Multicenter Clinical Study. Eur Urol. 2019 Apr;75(4):570-578. doi: 10.1016/j.eururo.2018.11.023. Epub 2018 Nov 23. PMID 30477981
- [Derived] Prive BM, Israel B, Schilham MGM, Muselaers CHJ, Zamecnik P, Mulders PFA, Witjes JA, Sedelaar M, Mehra N, Verzijlbergen F, Janssen MJR, Gotthardt M, Barentsz JO, van Oort IM, Nagarajah J. Evaluating F-18-PSMA-1007-PET in primary prostate cancer and comparing it to multi-parametric MRI and histopathology. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):423-430. doi: 10.1038/s41391-020-00292-2. Epub 2020 Sep 30. PMID 32999466